CLINICAL TRIAL: NCT03000959
Title: Stroke Unit in the Philippines: Is it Effective?
Brief Title: Stroke Unit in the Philippines: Is it Effective
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jose R. Reyes Memorial Medical Center (Other Government)
Responsible Party: Principal Investigator, Jose C. Navarro, Chairman Emeritus, Department of Neurology, Principal Investigator, Jose R. Reyes Memorial Medical Center
Other Study IDs: SU-PH1
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to assess the effectiveness of Stroke Unit in the Philippines by comparing the functional outcome between those patient admitted in the general neurology wards and stroke units using modified Rankin Scale

DETAILED DESCRIPTION:
This study aims to look into functionality of patient admitted in the stroke unit in the Philippines

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted in participating SUs starting June 2016 during acute stroke (within 7 days from onset), either hemorrhagic or ischemic stroke confirmed by CT-Scan or MRI, will be included

Exclusion Criteria:

* Patient who had previous of stroke and secondary cause of intracerebral hemorrhage such as trauma, arteriovenous malformation and aneurysm are not included in the study. Those who transferred from other institutions will be excluded. And also, patients who are below 18 years old are excluded in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients diagnosed with stroke (ischemic and hemorrhagic) starting on June 2016.
Sampling Method: Non-Probability Sample
Enrollment: 922 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | 3 Months

SECONDARY OUTCOMES:
Functional outcome in modified rankin scale | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Navarro, MD, Principal Investigator — Jose R. Reyes Memorial Medical Center
Locations (1):
- Jose R. Reyes Memorial Medical Center, Maño, Philippines

IPD SHARING:
Plan to Share IPD: Undecided
Computerized

REFERENCES:
- [Background] Langhorne P, de Villiers L, Pandian JD. Applicability of stroke-unit care to low-income and middle-income countries. Lancet Neurol. 2012 Apr;11(4):341-8. doi: 10.1016/S1474-4422(12)70024-8. Epub 2012 Mar 19. PMID 22441195
- [Background] Werner Hacke. The stroke care revolution. Lancet 2014; 383: 176-85
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Devuyst G, Bogousslavsky J. Clinical trial update: neuroprotection against acute ischaemic stroke. Curr Opin Neurol. 1999 Feb;12(1):73-9. doi: 10.1097/00019052-199902000-00012. PMID 10097888
- [Background] Peter Langhorne,Martin Dennis. Stroke Units: An evidence based approach. BMJ Books. 1998
- [Background] Counsell C, Warlow C, Sandercock P, Fraser H, van Gijn J. The Cochrane Collaboration Stroke Review Group. Meeting the need for systematic reviews in stroke care. Stroke. 1995 Mar;26(3):498-502. PMID 7886733
- [Background] Dennis MS, Langhorne P. Stroke Units: An evidence based approach. London, BMJ Publishing, 1998: Chapter 4, 33-40.
- [Background] The Stroke Society of the Philippines (SSP) Handbook of Stroke. 6th edition. 2014, 220-227.